CLINICAL TRIAL: NCT02383511
Title: A Phase 1b Placebo-controlled, Multi-centre, Randomized, Double-blind Dose Escalation Study to Evaluate the Pharmacokinetics (PK) and Safety of SMT C1100 in Patients With Duchenne Muscular Dystrophy (DMD) Who Follow a Balanced Diet
Brief Title: Modified Diet Trial: A Study of SMT C1100 in Paediatric Patients With DMD Who Follow a Balanced Diet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT C11003
Record Dates: First submitted 2015-02-04; First posted 2015-03-09 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — SMT C1100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sequence 1 (Other): Drug: SMT C1100 or placebo 3-treatment (Period 1,2 and 3)
  Interventions: Drug: SMT C1100
- Sequence 2 (Other): Drug: SMT C1100 or placebo 3-treatment (Period 1,2, and 3)
  Interventions: Drug: SMT C1100
- Sequence 3 (Other): Drug: SMT C1100 or placebo 3-treatment (Period 1,2 and 3)
  Interventions: Drug: SMT C1100

INTERVENTIONS:
Drug: SMT C1100 — Period 1, SMT C1100 1250 mg BID; Period 2, Placebo BID; Period 3, SMT C1100 2500 mg BID
  Arms: Sequence 1
Drug: SMT C1100 — Period 1, SMT C1100 1250 mg BID; Period 2, SMT C1100 2500 mg BID; Period 3, Placebo BID
  Arms: Sequence 2
Drug: SMT C1100 — Period 1, Placebo BID; Period 2, SMT C1100 1250 mg BID; Period 3, SMT C1100 2500 mg BID
  Arms: Sequence 3

SUMMARY:
Placebo-controlled, multi-centre, randomized, double-blind dose escalation study. The aim is to evaluate the pharmacokinetics (PK) and safety of SMT C1100 in paediatric patients with Duchenne Muscular Dystrophy (DMD) who follow a balanced diet.

DETAILED DESCRIPTION:
Primary Objective:

To determine the plasma concentration of SMT C1100 calculated at each time point for each subject (sample size (n), mean, standard deviation (SD), percentage of coefficient of variation (%CV), geometric mean, median, minimum, and maximum for the parent and the major metabolites).

Secondary Objectives:

1. To determine the safety and tolerability of single and multiple oral doses of SMT C1100 in patients with Duchenne Muscular Dystrophy (DMD) by assessing the participants adverse events, ECG results, vital signs and laboratory tests.
2. To evaluate the diurnal variability in the steady state PK of SMT C1100 calculated at each time point for each subject (sample size (n), mean, standard deviation (SD), percentage of coefficient of variation (%CV), geometric mean, median, minimum, and maximum for the parent and the major metabolites).
3. To evaluate reductions in creatine phosphokinase as a potential pharmacodynamic (PD) marker of SMT C1100 activity and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be males of any ethnic origin with a genetic diagnosis of DMD.
2. Children between 5 and 13 years of age.
3. A parent/legal guardian must date and sign a written consent on behalf of the patient, according to International Conference on Harmonisation (ICH) and local regulations. This person must understand the contents of the consent, requirements of the study and have had an opportunity to review questions with a medically trained member of the site study team.
4. The patient is willing to give verbal or written age appropriate assent to participate.
5. For safety reasons, the patient's parent/legal guardian must have a good understanding of the English language, which the consent/assent forms are available, and understand the requirements for reporting of any AE to the Investigator.
6. The patient has 6 months or more stable systemic (Patients using an intermittent regimen of steroid are allowed to be enrolled) corticosteroid therapy prior to Screening. Dose modifications for body weight are permitted.
7. The patient or parent is willing to adhere to a balanced diet from 1 week prior to dosing until the end of the follow-up period.
8. Patients must agree to not have sexual intercourse during the study treatment phases and until the end of their participation in the study.

Exclusion Criteria:

1. Enrolment or participation in any therapeutic clinical trial within the prior 3 months or 5 times the half-life (whichever is longer). Prior exposure to SMT C1100 is NOT an exclusion criterion.
2. Known hypersensitivity to the excipients of the study drug or a previous history of drug allergy.
3. The patient or parent is unwilling to adhere to a balanced diet from 1 week prior to dosing until the end of the follow-up period.
4. Is dairy or lactose intolerant, has an allergy to egg or nuts or any other dietary restrictions that might interfere with the conduct of the study.
5. Is unable to refrain from eating cruciferous vegetables and barbecued (chargrilled) meat for the duration of the study.
6. Use of prohibited medication within 5 half-lives prior to baseline assessments, unless otherwise stated in protocol.
7. Need for mechanical ventilation.
8. The patient experiences intermittent or continuous difficulties in swallowing.
9. Non ambulatory.
10. Any clinically significant acute illness within 4 weeks of the start of dose administration.
11. Any comorbidity that, in the opinion of the Investigator, increases the risk of participating in the study.
12. Symptomatic cardiomyopathy that in the opinion of the Investigator prohibits participation in this study.
13. Abnormality in the 12-lead ECG at the Screening visit that, in the opinion of the Investigator, increases the risk of participating in the study.
14. Any clinically significant medical condition, other than DMD that in the opinion of the Investigator may increase the risk of participating in the study or interfere with the interpretation of safety or efficacy evaluations (e.g., concomitant illness, severe reflux, psychiatric condition or behavioural disorder).
15. The Patient smokes or has exposure to daily passive smoking (including parent/legal guardian, siblings) so as to minimise environmental factors causing CYP 1A induction.
16. Excessive exercise (Investigator opinion).

Ages: 5 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters at different dose levels of SMT C1100 | 28 days
  To determine the plasma concentration of SMT C1100 parent and the major metabolites calculated at each time point for each subject.

SECONDARY OUTCOMES:
Safety and tolerability of SMT C1100 | 28 days
  To determine the safety and tolerability of single and multiple oral doses of SMT C1100 in patients with Duchenne Muscular Dystrophy (DMD) by assessing the participants adverse events.
Evaluation of plasma CK levels | 42 days
  To evaluate reductions in plasma creatine phosphokinase as a potential pharmacodynamic (PD) marker of SMT C1100 activity and muscle benefit.
Pharmacokinetic parameters at different dose levels of SMT C1100 | 28 Days
  To determine the plasma concentration of SMT C1100 major metabolites calculated at each time point for each subject.
Safety and tolerability of SMT C1100 | 28 Days
  To determine the safety and tolerability of single and multiple oral doses of SMT C1100 in patients with Duchenne Muscular Dystrophy (DMD) composite assessment of the participant's ECG results and laboratory tests.
Pharmacokinetic parameters at different dose levels of SMT C1100 | 28 Days
  To evaluate the diurnal variability in the steady state PK of SMT C1100 calculated at each time point for each subject.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Heart of England NHS Foundation Trust - Heart Lands Hospital, Birmingham
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust- Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Ricotti V, Spinty S, Roper H, Hughes I, Tejura B, Robinson N, Layton G, Davies K, Muntoni F, Tinsley J. Safety, Tolerability, and Pharmacokinetics of SMT C1100, a 2-Arylbenzoxazole Utrophin Modulator, following Single- and Multiple-Dose Administration to Pediatric Patients with Duchenne Muscular Dystrophy. PLoS One. 2016 Apr 7;11(4):e0152840. doi: 10.1371/journal.pone.0152840. eCollection 2016. PMID 27055247